CLINICAL TRIAL: NCT07183098
Title: A Prospective Observational Study on the Prevalence of Malnutrition and Clinical-Economic Aspects of the Impact of Specialized Nutritional Care on the 3-month Outcomes of Patients at High Risk of Malnutrition Admitted to a Rehabilitation Hospital
Brief Title: Prevalence and Clinical-Economic Aspects of Malnutrition in Rehabilitation
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: MalnutritionRehab_FDG
Record Dates: First submitted 2025-09-09; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Rehabilitation; Malnutrition
Keywords: Rehabilitation; Dietitians; Healthcare costs; MUST-Malnutrition Universal Screening Tool; malnutrition; Nutritional care
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participiants at high risk of malnutrition admitted to a rehabilitation hospital: Participiants at high risk of malnutrition who received standard nutritional care were compared with participiants at high risk of malnutrition who received specialized nutritional care
  Interventions: Other: Participiants at high risk of malnutrition who received standard nutritional care; Other: Participiants at high risk of malnutrition who received specialized nutritional care; Other: 3 month-post discharge evaluation

INTERVENTIONS:
Other: Participiants at high risk of malnutrition who received standard nutritional care — The overall clinical managment of people by ward's staff includes also nutritional care. Within 24-48 h after hospitalization, the ward's nursing staff screens people for nutritional risk using the Malnutrition Universal Screening Tool (MUST) tool. The attending ward's physician prescribes nutritional support and laboratory analyses in accordance with people's clinical needs and the underlying disease. Ward's physician cllinical judgement guides the decision to reassess and monitor the people's nutritional risk and status.
Other: Participiants at high risk of malnutrition who received specialized nutritional care — People referred to the Dietetic and Clinical Nutrition Service (DCNS) receive a structured, evidence-based diagnostic and therapeutic nutritional support. A dietitian performs a dietary assessment and the attending physicians of the DCNS prescribe a baseline set of laboratory analyses relevant for nutritional status. People referred to the DCNS are monitored regularly and systematically, daily or weekly according to the people's clinical condition and nutritional problems.
Other: 3 month-post discharge evaluation — Three months after discharge (follow-up), participiants of both groups were monitored through telephone interview to collect data regarding rate of hospital readmission, number of emergency department admissions, general practitioner visits, outpatient visits, diagnostic tests, daily medication use and survival.

SUMMARY:
The goal of this observational study is to learn about the clinical and economic aspects of specialized nutritional care in participiants at high risk of malnutrition (Malnutrition Universal Screening Tool-MUST equal or higher than 2) admitted to a rehabilitation hospital. The main questions it aim to answer are:

* Does a specialized nutritional care lower hospital readmission rate at three months post-discharge in participiants at high risk of malnutrition admitted to a rehabilitation hospital?
* Does a specialized nutritional care lower the number of emergency department admissions, number of general practitioner (GP) and outpatient visits, number of diagnostic tests and daily medication use and mortality rate in participiants at high risk of malnutrition admitted to a rehabilitation hospital?

Participiants at high risk of malnutrition, three months after discharge were monitored through telephone interview about the hospital readmission and mortality rate, the number of emergency department admissions, GP and outpatient visits, diagnostic tests and daily medication use for treatment burden.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the rehabilitation hospital IRCCS Fondazione Don Carlo Gnocchi ONLUS, Florence
* high risk of malnutrition (Malnutrition Universal Screening Tool-MUST equal or higher than 2)

Exclusion Criteria:

* age under 50 years;
* oncological diagnosis associated with a poor six-month prognosis and/or with advanced or irreversible cachexia;
* end-stage renal disease (dialysis);
* people already participating in a cardiac rehabilitation program at the time of enrollment;
* people with severe acquired brain injuries admitted for neurological rehabilitation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of people at high risk of malnutrition (Malnutrition Universal Screening Tool-MUST equal or higher than 2) admitted to the rehabilitation wards of the IRCCS Fondazione Don Carlo Gnocchi ONLUS.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital readmissions rate | 90 days post discharge
  The rate of hospital readmissions at three months post-discharge was computed as number of hospital readmissions from discharge to three-month follow-up.

SECONDARY OUTCOMES:
Emergency department admissions rate | 90 days post-discharge
  The rate of emergency department admissions was computed as the number of emergency department admissions from discharge to three-month follow-up.
General practitioner visits rate | 90 days post-discharge
  General practitioner visits rate was computed as the number of general practitioner visits from discharge to three-month follow-up
Outpatient visits rate | 90 days post-discharge
  The outpatient visits rate was computed as the number of outpatient visits from discharge to three-month follow-up
Diagnostic tests rate | 90 days post-discharge
  The diagnostic tests rate was computed as the number of diagnostic tests performed from discharge to three-month follow-up
Daily medication rate | 90 days post-discharge
  Daily medication rate is the number of drugs/day computed from discharge to three-month follow-up
Mortality rate | 90 days post-discharge
  Mortality rate was computed as the number of participiants dead from discharge to three-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa E Luisi, MD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi ONLUS
Locations (1):
- Fondazione Don Carlo Gnocchi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cederholm T, Bosaeus I, Barazzoni R, Bauer J, Van Gossum A, Klek S, Muscaritoli M, Nyulasi I, Ockenga J, Schneider SM, de van der Schueren MA, Singer P. Diagnostic criteria for malnutrition - An ESPEN Consensus Statement. Clin Nutr. 2015 Jun;34(3):335-40. doi: 10.1016/j.clnu.2015.03.001. Epub 2015 Mar 9. PMID 25799486
- [Background] Cederholm T, Barazzoni R, Austin P, Ballmer P, Biolo G, Bischoff SC, Compher C, Correia I, Higashiguchi T, Holst M, Jensen GL, Malone A, Muscaritoli M, Nyulasi I, Pirlich M, Rothenberg E, Schindler K, Schneider SM, de van der Schueren MA, Sieber C, Valentini L, Yu JC, Van Gossum A, Singer P. ESPEN guidelines on definitions and terminology of clinical nutrition. Clin Nutr. 2017 Feb;36(1):49-64. doi: 10.1016/j.clnu.2016.09.004. Epub 2016 Sep 14. PMID 27642056
- [Background] Cereda E, Lucchin L, Pedrolli C, D'Amicis A, Gentile MG, Battistini NC, Fusco MA, Palmo A, Muscaritoli M. Nutritional care routines in Italy: results from the PIMAI (Project: Iatrogenic MAlnutrition in Italy) study. Eur J Clin Nutr. 2010 Aug;64(8):894-8. doi: 10.1038/ejcn.2010.85. Epub 2010 May 26. PMID 20502467
- [Background] Lim SL, Ong KC, Chan YH, Loke WC, Ferguson M, Daniels L. Malnutrition and its impact on cost of hospitalization, length of stay, readmission and 3-year mortality. Clin Nutr. 2012 Jun;31(3):345-50. doi: 10.1016/j.clnu.2011.11.001. Epub 2011 Nov 26. PMID 22122869